CLINICAL TRIAL: NCT00147446
Title: Phase II Study of the Effects of Stress Management on Neuroimaging, Clinical, Immune and Psychosocial Outcomes
Brief Title: Stress Management for Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, David Mohr, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SIMS; R01HD043323 (NIH)
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Results first posted 2013-09-10 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Multiple Sclerosis
Keywords: Stress; Stress Management; Behavioral Medicine; Multiple Sclerosis; Psychoneuroimmunology
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individual Stress Management (Experimental): Stress management therapy for multiple sclerosis (SMT-MS) is a manualized, validated, published stress management program designed for patients with MS. Participants met with a therapist for 16 individual 50-minute sessions conducted over 20-24 weeks. The first 6 sessions focused on teaching problem solving skills, relaxation, increasing positive activities, cognitive restructuring, and enhancement of social support. Participants were able to tailor the treatment to meet their needs using optional treatment modules including communication and assertiveness training, fatigue management, anxiety reduction, pain management, management of cognitive problems, insomnia treatment, and management of sexual dysfunction.
  Interventions: Behavioral: Individual Stress Management
- Wait List Control (Other): Wait List Control provided treatment as usual for the first 10+ months of participation. A 5-hour workshop was provided after the 10th month. This allowed at least 2 post-treatment MRI evaluation that were not contaminated by the workshop.
  Interventions: Other: Wait List Control

INTERVENTIONS:
Behavioral: Individual Stress Management — Stress management therapy for multiple sclerosis (SMT-MS) is a manualized, validated, published stress management program designed for patients with MS. Participants met with a therapist for 16 individual 50-minute sessions conducted over 20-24 weeks. The first 6 sessions focused on teaching problem solving skills, relaxation, increasing positive activities, cognitive restructuring, and enhancement of social support. Participants were able to tailor the treatment to meet their needs using optional treatment modules including communication and assertiveness training, fatigue management, anxiety reduction, pain management, management of cognitive problems, insomnia treatment, and management of sexual dysfunction.
  Other Names: Cognitive Behavioral Stress Management for MS
  Arms: Individual Stress Management
Other: Wait List Control — Wait List Control provided treatment as usual for the first 10+ months of participation. A 5-hour workshop was provided after the 10th month. This allowed at least 2 post-treatment MRI evaluation that were not contaminated by the workshop.
  Arms: Wait List Control

SUMMARY:
There is a growing body of literature showing that stressful life events can increase the risk of developing exacerbations and new brain lesions among people with multiple sclerosis. The purpose of this study is to examine the hypothesis that stress management programs can reduce the occurrence of new brain lesions and exacerbations. We will also examine potential immune and neuroendocrine pathways.

DETAILED DESCRIPTION:
MS is a frequently disabling autoimmune disease affecting approximately 350,000 people in the United States. More than two decades of research has consistently shown a relationship between stressful life events (SLEs), in particular non-traumatic family and work stressors, and subsequent clinical exacerbation. Furthermore, we have shown that non-traumatic SLEs increase the risk of the subsequent appearance of new gadolinium enhancing (Gd+) magnetic resonance imaging (MRI) brain lesions, an early marker of MS inflammation and blood-brain barrier (BBB) breakdown. The purpose of this study is to determine the efficacy of cognitive behavioral stress management for MS (CBSM-MS) in reducing the occurrence of new brain lesions in people with relapsing forms of MS. Patients must have a documented new Gd+ MRI brain lesion or clinical exacerbation within the previous 12 months to be enrolled. One hundred and twelve patients will be enrolled for 12 months. Patients will be randomly assigned to either an intensive CBSM-MS program, consisting of 16 individual meetings with a behavioral medicine specialist, or a condensed CBSM-MS program, consisting of a one-day workshop offered after the 10th month of participation. Outcomes include MRI, clinical neurological end-points, and psychosocial functioning. We will also enhance our understanding of mechanisms by examining potential psychosocial, immune, and endocrine mediators of the relationship between SLEs and clinical and neuroimaging markers of MS inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MS
* New Gd+ MRI brain lesion or clinically diagnosed exacerbation within the previous 12 months.
* Able to speak english.
* Age 18 or over.
* Able to give informed consent.
* Patients taking the drug glatiramer acetate must have been on the drug for at least 6 months prior to their Gd+ MRI brain lesion and/or exacerbation.
* Patients taking an interferon beta drug must have been on the drug for at least 1 month prior to their Gd+ MRI brain lesion and/or exacerbation.
* Patients not on disease modifying treatment are not planning to initiate treatment.

Exclusion Criteria:

* Meets criteria for dementia by scoring below the 5th percentile in 3 or more of 6 areas of neuropsychological functioning or as determined by study neuropsychologist.
* Severe psychiatric pathology, including schizophrenia, bipolar disorder, current alcoholism or substance abuse, or other severe psychiatric disorder for which this intervention would be inappropriate.
* Active and severe suicidal ideation.
* Endocrine or metabolic disorder.
* Currently in psychotherapy.
* Initiated antidepressant therapy within the past 4 weeks.
* Received corticosteroid treatment within the past 28 days.
* Pregnant or planning pregnancy in the next 12 months.
* Has any non-removable metal or medical device in the body for which an MRI could pose a danger.
* Has any risk factors for developing nephrogenic systemic fibrosis (NSF) or is allergic to Gadolinium.
* Currently uses a Baclofen pump.
* Has an Expanded Disability Status Scale score greater than 6.5.
* Recently begun relaxation, meditation, yoga, or similar form of disease management course within the past 3 months.
* Treatment with Chemotherapy.
* Treatment with Tysabri.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2005-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C. Mohr, Ph.D., Principal Investigator — Northwestern University; Joyce Ho, PhD, Study Director — Northwestern University; David Daikh, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - UCSF Behavioral Medicine Research Center, San Francisco, California
  - Northwestern University, Department of Preventive Medicine, Chicago, Illinois
  - MS Center at Evergreen Medical Center, Kirkland, Washington

REFERENCES:
- [Background] Mohr DC, Lovera J, Brown T, Cohen B, Neylan T, Henry R, Siddique J, Jin L, Daikh D, Pelletier D. A randomized trial of stress management for the prevention of new brain lesions in MS. Neurology. 2012 Jul 31;79(5):412-9. doi: 10.1212/WNL.0b013e3182616ff9. Epub 2012 Jul 11. PMID 22786596
- [Derived] Burns MN, Nawacki E, Kwasny MJ, Pelletier D, Mohr DC. Do positive or negative stressful events predict the development of new brain lesions in people with multiple sclerosis? Psychol Med. 2014 Jan;44(2):349-59. doi: 10.1017/S0033291713000755. Epub 2013 May 17. PMID 23680407
- [Derived] Burns MN, Nawacki E, Siddique J, Pelletier D, Mohr DC. Prospective examination of anxiety and depression before and during confirmed and pseudoexacerbations in patients with multiple sclerosis. Psychosom Med. 2013 Jan;75(1):76-82. doi: 10.1097/PSY.0b013e3182757b2b. Epub 2012 Nov 28. PMID 23197840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at MS specialty clinics at three sites in the United States (University of California San Francisco California (UCSF), Evergreen Hospital Medical Center in Seattle Washington and the Feinberg School of Medicine at Northwestern University in Chicago Illinois) and through local chapters of the National MS Society.
Groups:
- Stress Management Therapy for Mulitple Sclerosis: Stress management therapy for MS(SMT-MS), provided 16 individual treatment sessions over 24 weeks, followed by a 24-week post-treatment follow-up.
- Wait List Control Condition: Wait list control provided treatment as usual for the first 10+ months of participants. A 5-hour workshop was provided afte the 10th month. This allowed at least 2 post-treatment MRI evaluations that were not contaminated by the workshop.
Period: Overall Study
Arm/Group | Stress Management Therapy for Mulitple Sclerosis | Wait List Control Condition
Started | 60 | 61
Completed | 60 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stress Management Therapy for Multiple Sclerosis: Stress management therapy for multiple sclerosis(SMT-MS)at baseline
- Wait List Control Condition: Wait list control provided treatment as usual for the first 10+ months of participation. A 5-hour workshop was provided after the 10th month. This allowed at least 2 post-treatment MRI evaluations that were not contaminated by the workshop
- Total: Total of all reporting groups
Arm/Group | Stress Management Therapy for Multiple Sclerosis | Wait List Control Condition | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 58 | 118
  >=65 years | 0 | 3 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 42.3 (9.03) | 43.0 (9.08) | 42.7 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 50 | 101
  Male | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  United States | 60 | 61 | 121

OUTCOME MEASURES:

1. Primary Outcome: No.of Gd+ Lesions From Week 8 to Week 24
Description: Gd+ is Gadolinium-enhancing MRI brain lesion, A marker of the opening of the blood-brain barrier and is typically used as a primary endpoints in phase II trials because of its high sensitivity to ongoing MS disease activity and its association with clinical exacerbation. The single value was calculated by summing up the lesions from week 8 to week 24.
Time Frame: week 8 to week 24
Population: A total of 121 patients with relapsing forms of MS were randomized to SMT-MS or WLC. Participants were enrolled at MS specialty clinics at 3 sites in the United States (UCSF; Evergreen Hospital Medical Center, and the Feinberg School of Medicine at Northwestern University, Chicago, Illinois) and through local chapters of the National MS Society.
Measure: Number; unit: participants
Groups:
- Stress Management Therapy for Multiple Sclerosis: Stress management therapy for MS(SMT-MS), provided 16 individual treatment sessions over 24 weeks, followed by a 24-week post-treatment follow-up.
- Wait List Control Condition: Wait list control(WLC) provided treatment as usual for the first 10+ months of participants. A 5-hour workshop was provided after the 10th month. This allowed at least 2 post-treatment MRI evaluations that were not contaminated by the workshop
Arm/Group | Stress Management Therapy for Multiple Sclerosis | Wait List Control Condition
Number analyzed (Participants) | 60 | 61
participants
  No. of Gd+ lesions(week 8 to week 24), Gd+ = 0 | 46 | 33
  No. of Gd+ lesions(week 8 to week 24), Gd+ = 1 | 5 | 13
  No. of Gd+ lesions(week 8 to week 24), Gd+ = 2 | 2 | 6
  No. of Gd+ lesions(week 8 to week 24), Gd+ = 3 | 2 | 6
  No. of Gd+ lesions(week 8 to week 24), Gd+ >= 4 | 5 | 3
Statistical Analysis 1: Comparison: Stress Management Therapy for Multiple Sclerosis vs Wait List Control Condition; It was hypothesized that treatment with stress management produced a significant reduction in cumulative Gd+ lesions compared to the control condition during the treatment period; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney); Wilcoxon two smaple test statistics = 2.09
Statistical Analysis 2: Comparison: Stress Management Therapy for Multiple Sclerosis vs Wait List Control Condition; It was hypothesized that significantly greater numbers of participants receiving stress management remained free of Gd+ lesions during the treatment, compared to those receiving the control condition; Test type: Superiority or Other; p = 0.02, Logistic Regression; Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.17 to 6.55]

2. Secondary Outcome: No.of New or Enlarged T2 Lesions From Week 8 to Week 24
Description: T2-weighted MRI is commonly used in phase II trials to identify more permanent lesions. The single value was calculated by summing up the lesions from week 8 to week 24.
Time Frame: week 8 to week 24
Measure: Number; unit: participants
Arm/Group | Stress Management Therapy for Mulitple Sclerosis | Wait List Control Condition
Number analyzed (Participants) | 60 | 61
participants
  No. of T2 lesions (week 8 to week 24), T2 = 0 | 43 | 26
  No. of T2 lesions(week 8 to week 24), T2 = 1 | 8 | 9
  No. of T2 lesions(week 8 to week 24), T2 = 2 | 1 | 9
  No. of T2 lesions(week 8 to week 24), T2 = 3 | 1 | 7
  No. of T2 lesions(week 8 to week 24), T2 >=4 | 7 | 10
Statistical Analysis 1: Comparison: Stress Management Therapy for Mulitple Sclerosis vs Wait List Control Condition; It was hypothesized that participants receiving SMT-MS showed a significant reduction in cumulative new T2 lesions, compared to those receiving the control condition during the treatment period; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney); Wilcoxon two sample test statistics = 2.84
Statistical Analysis 2: Comparison: Stress Management Therapy for Mulitple Sclerosis vs Wait List Control Condition; It was hypothesized that significantly greater numbers of participants receiving SMT-MS remained free of new T2 lesions during the treatment, compared to control condition participants; Test type: Superiority or Other; p = 0.006, Logistic Regression; Odds Ratio (OR) = 3.07, 95% CI 2-sided [1.38 to 6.81]

ADVERSE EVENTS:
Groups:
- Stress Management Therapy for Multiple Sclerosis: Stress management therapy for MS(SMT-MS, provided 16 individual treatment sessions over 24 weeks, followed by a 24-week post-treatment follow-up.
- Wait List Control Condition: Wait list control provided treatment as usual for the first 10+ months of participants. A 5-hour workshop was provided after the 10th month. This allowed at least 2 post-treatment MRI evaluations that were not contaminated by the workshop
Arm/Group | Stress Management Therapy for Multiple Sclerosis | Wait List Control Condition
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/61
Other Adverse Events (participants affected / at risk) | 0/60 | 0/61

LIMITATIONS AND CAVEATS:
we caution that it is premature to make specific clinical recommendations regarding the use of SMT-MS to manage MS disease-related activity. Future work should identify, refine, and optimize the active ingredients in this behavioral intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes